CLINICAL TRIAL: NCT02737787
Title: A Phase I Study of Concomitant WT1 Analog Peptide Vaccine or NY-ESO-1 Overlapping Peptides Vaccine in Combination With Nivolumab in Patients With Recurrent Ovarian Cancer Who Are in Second or Greater Remission
Brief Title: A Phase I Study of WT1 or NY-ESO-1 Vaccine and Nivolumab For Recurrent Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 15-247
Record Dates: First submitted 2016-04-05; First posted 2016-04-14 (Estimated); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Ovarian Cancer; Fallopian Tube; Primary Peritoneal Cancer; Recurrent Ovarian Cancer
Keywords: Second or Greater Remission; WT1 Analog Peptide Vaccine; NY-ESO-1 Overlapping Peptides; GM-CSF; Nivolumab; 15-247
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasm Metastasis | interventions — Nivolumab; NY-ESO-1-APH vaccine

STUDY DESIGN:
Intervention Model Description: This is an open-label, non-randomized phase I trial of a vaccine combined with anti-PD-1 (nivolumab) in patients with recurrent ovarian cancer who are in second or third clinical remission following additional chemotherapy.

ARMS (2):
- WT1 Vaccine and Nivolumab (Experimental): Patients will initially receive 6 vaccinations over 12 weeks and 7 infusions of nivolumab every two weeks over 14 weeks. Toxicity assessments will be performed with each dose of vaccine, and 3 weeks after the completion of therapy at week 15. Patients who do not have disease progression at the week 15 evaluation are permitted to receive 4 additional vaccines administered approximately every 8 weeks. This maintenance vaccine course would begin at week 19.This cohort has completed recruitment.
  Interventions: Biological: WT1 Vaccine; Drug: Nivolumab
- ESO-1 Vaccine and Nivolumab (Experimental): Patients will be vaccinated with the NY-ESO-1 OLP4 vaccine. Patients will receive a 1.0 mL emulsion of NY-ESO-1 OLPs with Poly-ICLC and Montanide.Nivolumab will be administered intravenously as a 30-minute infusion per institutional guidelines on weeks 0, 2, 4, 6, 8, 10 and 12.
  Interventions: Drug: Nivolumab; Biological: NY-ESO-1 Vaccine

INTERVENTIONS:
Biological: WT1 Vaccine
  Arms: WT1 Vaccine and Nivolumab
Drug: Nivolumab — Nivolumab will be administered intravenously as a 30-minute infusion per institutional guidelines on weeks 0, 2, 4, 6, 8, 10 and 12.
Biological: NY-ESO-1 Vaccine — Patients will be vaccinated with the NY-ESO-1 OLP4 vaccine. Patients will receive a 1.0 mL emulsion of NY-ESO-1 OLPs with Poly-ICLC and Montanide.
  Arms: ESO-1 Vaccine and Nivolumab

SUMMARY:
The purpose of this study is to test the safety of a combination of an investigational WT1 vaccine and another drug called nivolumab. This is the first time that the WT1 vaccine and nivolumab are being used in combination. Also, to test the safety of a combination of an investigational NY-ESO-1 vaccine and another drug called nivolumab.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of ovarian, fallopian tube or primary peritoneal cancer confirmed by pathology review at MSK.
* Patients will have relapsed at least once and returned to complete clinical remission after additional chemotherapy. Interval surgery is permitted.
* Complete clinical remission is defined as CA-125 within normal limits, examination and CT or MRI without objective evidence of disease (non specific abnormalities are permitted on radiologic imaging).
* Patients may sign screening consent during recurrence or at time of remission if they can start vaccine therapy within 4 months of completing chemotherapy.
* Testing of patient's archived (paraffin embedded, unstained slides) or freshly biopsied tumor nodules must be positive for WT1 (Cohort 1) or NY-ESO-1 (Cohort 2) protein expression. WT1 expression: Immunohistochemical analysis will be performed using the technique described by Dupont et al [58]. WT1 expression will be graded according to an adaptation of the German Immunoreactive Score (IRS). Only tumors with moderate to strong IRS scores (4-12) will be considered WT1 positive.
* NY-ESO-1 expression: Tissue available from primary and/or recurrent disease will be evaluated for tumor expression of NY-ESO-1 by immunohistochemical (IHC) and/or RT-PCR analysis will be performed using the technique described by Jungbluth et al
* Age ≥ 18 years
* Karnofsky performance status ≥ 70%
* Hematologic parameters: Absolute neutrophil count ≥ 1000/mcL, Platelets > 50 K/mcL.
* Biochemical parameters: Total bilirubin ≤ 1.5 mg/dl, AST and ALT ≤ 2.5 x upper limits of normal, Creatinine ≤ 1.5 mg/dl.
* Patient of childbearing potential must have a negative serum pregnancy test prior to study entry and must be practicing and effective form of birth control

Exclusion Criteria:

* Pregnant or lactating women
* Patients with active infection requiring systemic antibiotics, antiviral, or antifungal treatments
* Patients with a serious unstable medical illness or another active cancer.
* Patients with a condition requiring systemic treatment with either corticosteroids (>10mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses >10mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Patients with known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Patients with known active hepatitis B virus or hepatitis C virus acute or chronic infection.
* Patients with active known or suspected autoimmune disease (treated hypothyroidism is permitted to enroll)
* Patients with active interstitial pneumonitis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 30 days
  The first 3 patients will be observed for 30 days before enrolling the next 7 patients. Accrual will continue as patients become available after the first 3 patients are observed for 30 days. If >2/10 DLTs are observed then the study combination will not be considered safe.

SECONDARY OUTCOMES:
immune response (cohort 2) | week 15
  Serologic IgM and IgG antibody responses will be measured by ELISA against each antigen
progression-free survival rate (cohort 2) | 1 year
  Will evaluate PFS rate at 1-year using Kaplan Meier methodology

CONTACTS AND LOCATIONS:
Overall Officials: Roisin O'Cearbhaill, MB BCh BAO, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All protocol activities), Rockville Centre, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/